CLINICAL TRIAL: NCT02193672
Title: A Pilot, Exploratory, Non-Randomized Study of PET/CT With the Investigational Agent [18F] Fluciclatide to Correlate With Response to Anti-Cancer Therapy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-0591
Record Dates: First submitted 2014-07-11; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Cancers
Keywords: Advanced cancers; PET/CT; Positron emission tomography / computed tomography; [18F]Fluciclatide; Chemotherapy; Phone calls
MeSH Terms: interventions — AH 111585; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET/CT + [18F]Fluciclatide (Experimental): At baseline: Participants have PET/CT imaging within 7 days prior to initiation of chemotherapy treatment. Participants monitored at 24 hours post scan via telephone.
  On treatment: Participants have PET/CT imaging at end of the first cycle and prior to the initiation of the second cycle of chemotherapy. Participants assessed at 24 hours post scan via telephone call.
  Baseline and on treatment PET/CT imaging performed with agent [18F] Fluciclatide.
  Interventions: Drug: [18F] Fluciclatide; Procedure: PET/CT Scan; Behavioral: Phone Calls

INTERVENTIONS:
Drug: [18F] Fluciclatide — [18F] Fluciclatide given by vein before PET/CT scan.
Procedure: PET/CT Scan — PET/CT scan performed at treatment baseline visit, and about 1 week before first cycle of chemotherapy. Then, a PET/CT scan performed at end of first cycle of chemotherapy.
  Other Names: Positron emission tomography / computed tomography
Behavioral: Phone Calls — Phone call to participants by study staff about 24 hours after each PET/CT is performed.

SUMMARY:
The goal of this clinical research study is to find out if using the tracer (liquid used in imaging scans) [18F]fluciclatide in positron emission tomography / computed tomography (PET/CT) scans will help researchers learn more quickly if the disease is responding to treatment.

DETAILED DESCRIPTION:
PET/CT Scans:

If you are found eligible to take part in this study, you will have a PET/CT scan at your treatment baseline visit, about 1 week before your first cycle of chemotherapy. You will then have a second PET/CT scan at the end of your first cycle of chemotherapy (about 3-4 weeks after starting chemotherapy).

For up to 6 hours before the PET/CT scan, you must not eat or drink anything except water. A small needle and tube will be placed in your arm, and you will receive an injection of a very small amount of a mildly radioactive material into your bloodstream (the investigational tracer, [18F]fluciclatide). The radioactive nature of this injected material allows the scanner to "see" it in certain places in your body. After the injection, you will need to rest quietly until it is time for the scan. The amount of rest time may vary, but be prepared to wait for between 45 and 90 minutes. During the scan, you will lie flat on your back on a table. The scan itself may last up to 1 hour.

Each PET/CT imaging session will last about 4 hours total from the time you arrive at the clinic until you are discharged and allowed to go home. You may be discharged 30 minutes after the scan is complete, if the doctor thinks you are clinically stable and it is safe for you to leave.

Study Visits:

If the following tests are already being performed as part of the clinical research study you are participating in or as part of standard care, they will not need to be repeated for this study.

Baseline Visit (before the first PET/CT is performed):

* You will have a physical exam.
* Blood (about 3 tablespoons) will be drawn for routine tests.
* If you can become pregnant, urine will be collected for a pregnancy test. To take part in this study, you must not be pregnant.

End of Cycle 1 (before the second PET/CT is performed):

-Blood (about 3 tablespoons) will be drawn for routine tests.

About 24 hours after each PET/CT is performed, the study staff will call you by telephone to ask about your health status and any side effects you may be experiencing.

Anytime within the next month after the second PET/CT scan, blood (about 3 tablespoons) will be drawn for routine tests.

When your chemotherapy is over, you will have a third PET/CT scan as part of your standard care, and an FDG tracer will be used for that scan.

Length of Participation:

Your study participation will end about 6 weeks after your second PET/CT scan is performed.

This is an investigational study. [18F]Fluciclatide is not FDA approved or commercially available. At this time, it is only being used in research.

Up to 50 patients will take part in this research study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is >/= 18 years and male or female of any race/ethnicity.
2. Patient or patient's legally authorized representative provides written informed consent and is willing to comply with protocol requirements.
3. Patient must be scheduled to receive an anti-VEGF inhibitor (bevacizumab, sorafenib, sunitinib, other), mTOR inhibitor (temsirolimus, everolimus, other), or other molecules with antiangiogenic properties including taxol as anti-cancer therapy.
4. Patient must have normal hepatic and renal function defined as: 1) AST (SGOT)/ALT (SGPT) </=3 x institutional upper limit of normal and 2) serum creatinine </= 2x institutional upper limit of normal.
5. Platelet count of > 75 x 10^3/μL
6. Patients may participate in clinical trials in the Phase I program.
7. Patients with any solid tumor type.

Exclusion Criteria:

1. Patient is not capable of complying with study procedures.
2. Female patient is pregnant or nursing; exclude the possibility of pregnancy by one of the following: 1) Confirming in medical history that the patient is postmenopausal defined as 12 consecutive months of amenorrhea, or surgically sterile, 2) Confirming the patient is using one of the following methods of birth control for a minimum of one month prior to entry into this study: Intrauterine device (IUD), oral contraceptives, Depo-Provera, or Norplant, 3) Confirming a negative urine dipstick test taken the morning of receiving the investigational agent [18F]fluciclatide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in Tumor Uptake | After 2, four week chemotherapy cycles
  Primary efficacy endpoint is change in tumor uptake of investigational agent [18F]Fluciclatide, as measured by standardized uptake value (SUVFluciclatide) from before treatment to after one cycle of treatment but before the second cycle starts. This determined from investigational agent [18F]Fluciclatide PET scans. Changes in SUVFluciclatide compared to standard tumor's response measured after completion of 2 cycles of treatment as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) as well as tumor size change as a continuous variable measured by the standard CT or PET/CT scans. Tumor size can also be measured by the WHO two-dimensional measurement in addition to the Response Evaluation Criteria in Solid Tumors (RECIST), one-dimensional measurement. Changes in SUVFluciclatide after one cycle also compared to tumor volume and tumor size as continuous variables after two cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolia M. Tsimberidou, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org